CLINICAL TRIAL: NCT03883737
Title: Effect of the Ultrasound-guided Percutaneous Neuromodulation on the Anterior Pain Knee: a Pilot Study
Brief Title: Percutaneous Neuromodulation on the Anterior Pain Knee
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Seville (Other)
Responsible Party: Principal Investigator, Blanca de la Cruz Torres, Director, University of Seville
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: PNM and knee
Record Dates: First submitted 2019-03-16; First posted 2019-03-21 (Actual); Last update posted 2020-07-14 (Actual); Status verified 2020-07

CONDITIONS: Neuromodulation; Anterior Pain Knee; Femoral Nerve

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group 1: PNM in pain knee (Experimental): participants in whom PNM will be applied to the femoral nerve of the pain knee
  Interventions: Other: PNM
- Group 2: PNM in non-pain knee (Experimental): participants in whom PNM will be applied to the femoral nerve of the non-pain knee
  Interventions: Other: PNM

INTERVENTIONS:
Other: PNM — an asymmetric rectangular biphasic current (250 microseconds, 10 Hz)

SUMMARY:
Anterior knee pain (AKP) is one of the most frequent pathologies of the lower limb, in young and adult subjects. In the field of Physiotherapy, ultrasound-guided Percutaneous Neuromodulation (PNM) is defined as the application through a needle with ultrasound guidance of an electrical current at low or medium frequency, seeking a sensitive and / or motor response of a peripheral nerve in some point of its trajectory, or of a muscle in a motor point, with a therapeutic objective. The objective of this study is to analyze that the effect of PNM on the femoral nerve produces statistically significant changes in pain, joint range and knee functionality in patients with chronic AKP. Thirty subjects will be recruited, which will be divided into 2 groups: group 1 to which PNM will be applied to the femoral nerve of the pain knee; and group 2 to which PNM will be applied to the femoral nerve of the non-pain knee. The PNM intervention with NMP will consist in the single application of an asymmetric rectangular biphasic current (250 microseconds, 10 Hz)

ELIGIBILITY:
Inclusion Criteria:

* chronic anterior knee pain >3 months
* older than 18 years-old

Exclusion Criteria:

* Surgical intervention in the intervention area
* Prosthesis or osteosynthesis in the intervention area
* Cardiac or tumoral diseases
* Coagulopathies
* Be under the effects of certain medications
* contraindication characteristic of the puncture

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 28 (Actual)
Dates: Start 2019-04-14 (Actual); Primary Completion 2019-04-15 (Actual); Study Completion 2019-11-01 (Actual)

PRIMARY OUTCOMES:
visual analog scale (VAS) (0, no pain; 100, maximum pain). | up to 1 week
  pain
range joint | up to 1 week
  goniometer
VISA-p questionnaire (0, maximum pain; 100, no pain). | up to 1 week
  Functional pain
Kujala questionnaire (0, maximum pain; 100, no pain). | up to 1 week
  Functional pain

CONTACTS AND LOCATIONS:
Locations (1):
- University of Seville, Seville, Spain